CLINICAL TRIAL: NCT07280793
Title: Visualizing CAR-T Cell Therapy in Multiple Myeloma Using a BCMA-Targeted PET Probe
Brief Title: CAR-T Cell Efficacy With Molecular Imaging in Multiple Myeloma
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Xuzhou Medical University (Other)
Responsible Party: Principal Investigator, Kai Lin Xu，MD, Chief physician, Xuzhou Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XYFY2025-KL519-01
Record Dates: First submitted 2025-11-17; First posted 2025-12-12 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Non-invasive CAR-T Cell Monitoring; BCMA-targeted PET Imaging; CAR-T Cell Biodistribution and Persistence; GMP-compliant Radiopharmaceutical Preparation
Keywords: ⁶⁸Ga-NOTA-BCMA; BCMA CAR-T cell imaging; BCMA PET tracer; Radiolabeled BCMA peptide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 68Ga-NOTA-BCMA (Experimental): Eligible subjects enrolled in the study will receive a predetermined dose of the 68Ga-NOTA-BCMA radiopharmaceutical preparation as part of the investigational imaging protocol.
  Interventions: Other: BCMA-Targeting CAR-T Cell Therapy; Device: PET/CT Imaging

INTERVENTIONS:
Other: BCMA-Targeting CAR-T Cell Therapy — Patient T-cells are harvested and genetically engineered to express chimeric antigen receptors (CARs) targeting B-cell maturation antigen (BCMA). These modified CAR-T cells specifically recognize and eliminate multiple myeloma cells expressing BCMA. Following reinfusion, the CAR-T cells undergo antigen-stimulated proliferation, establishing sustained antitumor immune activity.
Device: PET/CT Imaging — A low-dose PET/CT scan will be performed 60 minutes post-administration of the agent. Low-dose CT is only utilized for anatomic localization and PET attenuation correction, and the radiation dose involved is substantially lower than that of conventional CT.

SUMMARY:
⁶⁸Ga-NOTA-BCMA is a novel, targeted PET tracer under clinical investigation. It is designed to provide a non-invasive method for monitoring the biodistribution and persistence of BCMA CAR-T cells in patients. Preclinical data robustly support its specific binding, favorable pharmacokinetics, and excellent safety profile, warranting its advancement into clinical studies.

DETAILED DESCRIPTION:
⁶⁸Ga-NOTA-BCMA is an investigational PET radiopharmaceutical designed for targeted in vivo tracking of BCMA-directed CAR-T cells. Its molecular design incorporates a BCMA-derived peptide, specific for the CAR's scFv, conjugated to the ⁶⁸Ga-chelator NOTA. Preclinical data confirm high target affinity, rapid renal clearance (t₁/₂α=3.30 min, t₁/₂β=33.27 min), and an excellent safety profile with no drug-related toxicities in murine models. The agent is administered as a single IV bolus (4 mCi/80 μg) and must be used within 4 hours of GMP-compliant, on-site radiolabeling.

ELIGIBILITY:
Inclusion Criteria:

* **Inclusion Criteria**

  1. Subjects must voluntarily sign the informed consent form and be able to complete the trial per the protocol requirements.
  2. Age 18 years or older, regardless of gender.
  3. Diagnosed with multiple myeloma and scheduled to receive anti-BCMA CAR-T cell therapy.
  4. ECOG performance status of 0-2; with a life expectancy of not less than 3 months.
  5. Female subjects of childbearing potential must have a negative serum pregnancy test prior to enrollment.
  6. For female subjects of childbearing potential or male subjects with partners of childbearing potential, agreement to remain abstinent or use one or more forms of contraception with a failure rate of <1% per year during the study period and for at least one year after the study completion.

Exclusion Criteria:

* **Exclusion Criteria**

  1. Participation in another interventional clinical trial, concurrently or within 28 days prior to the first dose in this study. Participation in non-interventional trials is permitted.
  2. History of hypersensitivity to any component of the imaging agent or antibodies, or a known allergic predisposition.
  3. Inability to undergo PET/CT imaging, such as due to claustrophobia or emotional instability.
  4. Current use of anticoagulant therapy or anticipated requirement for such therapy during the study period.
  5. Known allergic or hypersensitivity reactions to biological products or any excipient of the 68Ga-NOTA-BCMA molecular probe.
  6. Active hepatitis B or C infection, or seropositivity for human immunodeficiency virus (HIV) antibody or Treponema pallidum antibody.
  7. Pregnancy, lactation, or intention to become pregnant during the trial period.
  8. Any other condition deemed by the investigator to render the subject unsuitable for trial participation.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-12-17 (Estimated); Primary Completion 2027-12-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Biodistribution of 68Ga-NOTA-BCMA | Baseline (pre-CAR-T), and at Day 6±2, Day 11±2, Day 21±2 post-CAR-T infusion (Scan at 60 minutes post-injection). For the first 3 subjects, additional scans at 30 and 120 minutes post-injection will be performed at baseline.
  Assessment of tracer uptake in tumor and normal tissues (e.g., brain, liver, heart) by measuring Standardized Uptake Values (SUV) on low-dose PET/CT scans.
Pharmacokinetic assessment of 68Ga-NOTA-BCMA: measurement of elimination half-life (t1/2) | Baseline: pre-injection, and at 2, 5, 10, 15, 30, 60, 90, 120 minutes post-injection of 68Ga-NOTA-BCMA. (May be omitted for subsequent subjects based on results from the first 5 subjects).
  Measure the elimination half-lives of radioactive concentrations in whole blood and plasma at multiple time points to characterize the clearance kinetics of the tracer.

SECONDARY OUTCOMES:
CAR-T Cell Expansion and Persistence | Day 6±2 and Day 11±2 post-CAR-T infusion.
  Quantitative measurement of CAR-T copy number in peripheral blood using qPCR.
Safety and Tolerability of 68Ga-NOTA-BCMA | Vital signs: pre-injection and 2 hours (±1h) post-injection of 68Ga-NOTA-BCMA. Other safety assessments: throughout the study, with a follow-up at Day 28±2 after the last tracer dose.
  The number of participants with adverse events is assessed via the NCI Common Terminology Criteria for Adverse Events (CTCAE) V5.0.
  The number of participants with abnormal vital signs is assessed using electronic thermometers, electronic sphygmomanometers, electronic monitors (for heart rate), and manual chest rise counting.
  The number of participants with abnormal physical examination findings is assessed in accordance with standard clinical protocols.
  The number of participants with laboratory abnormalities (including hematology, urinalysis, coagulation, and blood biochemistry) is assessed using automated analyzers (for hematology, coagulation, and blood biochemistry), dry chemistry analyzers, and sediment microscopes (for urinalysis).
  The number of participants with abnormal electrocardiogram (ECG) findings is assessed via 12-lead electrocardiograph testing.
CAR-T Cell Immunophenotyping | Day 6±2 and Day 11±2 post-CAR-T infusion.
  Characterization of CAR-T cell populations in peripheral blood using flow cytometry.

CONTACTS AND LOCATIONS:
Overall Officials: Xueyan Zhou, M.D., Ph.D., Principal Investigator — Xuzhou Medical University

IPD SHARING:
Plan to Share IPD: No